CLINICAL TRIAL: NCT00745173
Title: An Open-Label, Single/Multiple Dose Non-Randomized, 3-Period, Crossover Study To Determine The Potential Drug Interaction Of Conjugated Estrogens (CE) On Bazedoxifene In Healthy Postmenopausal Women.
Brief Title: Study Evaluating Premarin and Bazedoxifene Potential Interaction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3115A1-1135
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Postmenopause
MeSH Terms: interventions — Estrogens, Conjugated (USP)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: Premarin

INTERVENTIONS:
Drug: Premarin

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (absorption, distribution, breakdown and elimination in the body) of a single dose of bazedoxifene (BZA) 20 mg tablet when administered together with multiple doses of Premarin (conjugated estrogens or CE) to healthy postmenopausal women.

Information will also be obtained regarding the safety and tolerability of this combination in healthy, postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion into the study, women must be healthy and postmenopausal (either naturally or surgically) between the ages of 35 and 70, inclusive.
* Blood hormone levels must be consistent with a postmenopausal state (for specified subjects).
* They can either be a non-smoker or smoke less than 10 cigarettes per day, and be able to abstain from smoking during clinic confinements

Exclusion Criteria:

* A subject will be excluded from participation if they :
* Have participated in a clinical drug study within 30 days prior to study medication administration;
* Have a history of drug or alcohol abuse within 1 year or consume more than 2 standard units per day of alcohol (a standard unit equals 12 ounces of beer, 1 ½ ounces of 80-proof alcohol or 6 ounces of wine);
* Donate any other plasma or blood during the total study.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (absorption, distribution, breakdown and elimination in the body) parameters | 3 months

SECONDARY OUTCOMES:
To continue assessment of the safety profile as well as the tolerability the two drugs administered in combination in this population. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Dr. David Carter, Austin, Texas, United States